CLINICAL TRIAL: NCT00070850
Title: The Feasibility of Screening for Smith-Lemli-Opitz Syndrome
Brief Title: Prenatal Screening For Smith-Lemli-Opitz Syndrome
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: R01HD038940 (NIH)
Record Dates: First submitted 2003-10-08; First posted 2003-10-13 (Estimated); Last update posted 2007-07-02 (Estimated); Status verified 2005-08

CONDITIONS: Smith-Lemli-Opitz Syndrome; Pregnancy
Keywords: Screening; Prenatal; Amniocentesis
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Smith-Lemli-Opitz Syndrome (SLOS) is a genetic condition that causes mental retardation and other birth defects. This study will evaluate a new prenatal screening test for SLOS.

DETAILED DESCRIPTION:
SLOS is an inherited metabolic disorder characterized by moderate to severe mental retardation and congenital anomalies. SLOS is caused by a deficiency of the enzyme 7-dehydrocholesterol reductase and the resulting defect in the conversion of 7-dehydrocholesterol to cholesterol. SLOS can now be reliably detected prenatally by analysis of amniotic fluid 7-8- dehydrocholesterol (7/8-DHC) levels. Unconjugated estriol (uE3) is one of the maternal serum analytes currently measured routinely to screen for Down syndrome. This analyte requires cholesterol as a precursor, and its concentration in maternal serum is lower when the fetus has SLOS.

Currently, there is no national standard for the approach taken in prenatal screening; existing programs vary both in availability and in the protocol and algorithms used. The major barrier to identifying SLOS prenatally is the absence of sound screening methodology that takes into account the detection rate, the false positive rate, and the prevalence. This study will evaluate the efficacy of routinely identifying Smith-Lemli-Opitz Syndrome (SLOS) prenatally.

The screening model in this study is based on data from SLOS pregnancies and will be tested in 1,000,000 pregnancies in which maternal serum uE3, alpha-fetoprotein, and human chorionic gonadotrophin measurements are being done as part of routine screening for Down syndrome. The screening false positive rate is projected to be 0.34%, the detection rate 62%, and the odds of being affected given a positive screening result 1:70. These rates all compare favorably with prenatal screening tests now in routine use. The study will also determine whether SLOS diagnostic studies can be carried out in maternal urine or serum, rather than amniotic fluid, thereby avoiding invasive procedures.

Participants in this study will be pregnant women undergoing amnioscentisis during the second trimester. Women who have a positive test for SLOS will be asked to provide a urine and blood sample. The study will collect data on patient demographics and family history; data will also be obtained from the participant's ultrasound, karyotype, alpha-fetoprotein, maternal serum screening, and SLOS reports. Three months after the pregnancy due date, a genetic counselor will contact the participant to obtain basic information about the baby's delivery and health.

ELIGIBILITY:
Inclusion Criteria

* Pregnant, second trimester
* Singleton pregnancy
* Positive second trimester maternal serum screen for Smith-Lemli-Opitz Syndrome (using the Foundation for Blood Research screening algorithm )

Exclusion criteria:

* Gestational age at time of serum collection outside the range accepted for Down Syndrome screening
* Not pregnant
* Twin/multiple pregnancy
* Sample/clerical/assay error
* Physician not participating in study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1800
Dates: Start 2001-04; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: James E. Haddow, M.D., Principal Investigator — Foundation for Blood Research
Locations (1):
- Foundation for Blood Research, Scarborough, Maine, United States

REFERENCES:
- [Background] Palomaki GE, Bradley LA, Knight GJ, Craig WY, Haddow JE. Assigning risk for Smith-Lemli-Opitz syndrome as part of 2nd trimester screening for Down's syndrome. J Med Screen. 2002;9(1):43-4. doi: 10.1136/jms.9.1.43. PMID 11943798